CLINICAL TRIAL: NCT00961207
Title: Study of Triple Blockade of the Renin Angiotensin Aldosterone System (RAAS) in Diabetic (Type 1&2) Proteinuric Patients With (ACE-, ARB, DRI)
Brief Title: Triple Blockade of the Renin Angiotensin Aldosterone System in Diabetic (Type 1&2) Proteinuric Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Altitude trial which used similar drugs was terminated due to increased ADR.
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Pete Antonopoulos, Clinical Pharmacist, Cook County Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHStrogerH09-083
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Microalbuminuria; Macroalbuminuric Diabetic Nephropathy; Diabetes; Proteinuria; Albuminuria
MeSH Terms: conditions — Diabetes Mellitus; Proteinuria; Albuminuria | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren in Macroalbuminuria (Active Comparator): Aliskiren 150 mg daily for 2 weeks and then increased to 300 mg daily for 4 weeks.
  Interventions: Drug: Aliskiren
- Aliskiren Microalbuminuria (Active Comparator): Aliskiren 150 mg daily for 2 weeks and then increased to 300mg daily for 4 weeks
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150mg daily for 2 weeks and increased to 300 mg daily for 4 weeks.
  Other Names: Tekturna
  Arms: Aliskiren in Macroalbuminuria
Drug: Aliskiren — Aliskiren 150mg daily for 2 weeks and increased to 300 mg daily for 4 weeks.
  Other Names: Tekturna
  Arms: Aliskiren Microalbuminuria

SUMMARY:
Study Hypothesis:

Reduction in albuminuria has been shown to decrease progression of diabetic

nephropathy. In diabetic nephropathy patients treated with maximal

antihypertensive doses with dual RAAS blockade (total daily dose valsartan 320

mg and either enalapril 40 mg or benazepril 40 mg daily, or losartan 100mg), persistent

albuminuria reflects further additional RAAS activation. Microvascular renal

disease due to increased RAAS activation may be more effectively treated with

triple blockade by the addition of a direct renin inhibitor (DRI) Aliskiren.

ELIGIBILITY:
Inclusion Criteria:

* Macroalbuminuria > 300mg/g
* Microalbuminuria 30-300mg/g
* Stable on max dose of an ACE-I or ARB (Can also be titrated to max dosage of ACE-I and ARB and stable on those doses for at least 2 weeks)
* Blood pressure <130/80 mm Hg at time of enrollment
* Diabetic either Type 1 or 2

Exclusion Criteria:

* GFR <60 m/min
* Potassium > 5mg/dl at time of enrollment
* Pregnant
* History of Angioedema
* ACE-I cough
* Allergic to ARB, ACE-I, DRI
* A1C > 9%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduction in albuminuria/proteinuria | 6 weeks

SECONDARY OUTCOMES:
Safety of Triple RAAS inhibition with ACE-I, ARB and DRI | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pete Antonopoulos, PharmD, Principal Investigator — Cook County Health
Locations (1):
- John H Stroger Hospital of Cook County, Chicago, Illinois, United States